CLINICAL TRIAL: NCT01486966
Title: A 2-week, Randomised, Controlled, Open-label, Two-group Parallel, Multi-centre Trial Comparing Efficacy and Safety of Insulin Detemir Plus Insulin Aspart and NPH Insulin Plus Human Soluble Insulin Both in a Basal Bolus Regimen With or Without Metformin in Chinese Inpatients With Type 2 Diabetes Currently Treated With Insulin Qualifying for Intensified Treatment
Brief Title: Comparing Efficacy and Safety of Insulin Detemir Plus Insulin Aspart and NPH Insulin Plus Human Soluble Insulin With or Without Metformin in Chinese Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Trial terminated prematurely due to slow recruitment.
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-3954; U1111-1123-7088 (Other: WHO)
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Aspart; Insulin, Isophane; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin detemir / IAsp (Experimental)
  Interventions: Drug: insulin detemir; Drug: insulin aspart; Drug: metformin
- insulin NPH (Active Comparator)
  Interventions: Drug: insulin NPH; Drug: human soluble insulin; Drug: metformin

INTERVENTIONS:
Drug: insulin detemir — Dose individually adjusted. Administered subcutaneously/s.c. (under the skin) once daily using NovoPen®4
  Arms: Insulin detemir / IAsp
Drug: insulin aspart — Dose individually adjusted. Administered subcutaneously/s.c. (under the skin) three times a day before a meal using NovoPen®4
  Arms: Insulin detemir / IAsp
Drug: insulin NPH — Dose individually adjusted. Administered subcutaneously/s.c. (under the skin) once daily using NovoPen®4
  Arms: insulin NPH
Drug: human soluble insulin — Dose individually adjusted. Administered subcutaneously/s.c. (under the skin) three times a day before a meal using NovoPen®4
  Arms: insulin NPH
Drug: metformin — For subjects previously treated with metformin, the dosage and frequency will be kept unchanged

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to compare efficacy and safety of insulin detemir plus insulin aspart and NPH insulin plus human soluble insulin both in a basal bolus regimen with or without metformin in Chinese patients with type 2 diabetes.

The trial adopts a group sequential design, where the analysis of the primary efficacy endpoint will be performed at the interim analysis, in addition to the final formal analysis. The decision to continue or stop the trial will be based on the result of the interim analysis.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed clinically) for at 12 months or longer
* Currently treated with basal insulin once daily or premixed insulin twice daily for at least 3 months with or without OAD(s), and total daily insulin dose less than 1.4 IU (U)/kg (If treated with metformin, unchanged total daily dose of at least 1000 mg for at least 3 months)
* Body Mass Index (BMI) equal to 40 kg/m^2 or below
* HbA1c (glycosylated haemoglobin A1c) between 7.0% and 10.0% by central laboratory analysis
* Plan to be admitted for optimising glycaemic control at least 2 days prior to the randomisation

Exclusion Criteria:

* Treatment with thiazolidinediones (TZD) or Glucagon-Like Peptide-1 (GLP-1) receptor agonists within the last 3 months prior to the screening
* Anticipated change after the randomisation in concomitant medication known to interfere with glucose metabolism, such as systemic corticosteroids, beta-blockers and mono amine oxidase (MAO) inhibitors
* Previous participation in this trial (participation is defined as randomised. Re-screening of screening failures is allowed only once within the limits of the recruitment period.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- China (5):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Wuxi, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality

REFERENCES:
- [Result] Guo X, Li Q, Shi Y, Bu R, Liu J, Qu S, Gao Y. Efficacy and safety of insulin detemir plus insulin aspart versus NPH insulin plus human soluble insulin with or without metformin in Chinese type 2 diabetes. Chinese J Diabetes 2014; 22 (1)
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6 centres in China participated.
Pre-assignment Details: Between screening and treatment with trial drugs, subjects were assessed for eligibility and were randomised 1:1 into one of the two treatment arms.
Groups:
- Insulin Detemir + Insulin Aspart ± Metformin: Insulin detemir was administered subcutaneously in the thigh once daily at bedtime as basal insulin. Insulin aspart was injected in the abdominal area subcutaneously 0~5 minutes before each meal as bolus insulin. Metformin was given to subjects who were taking metformin before this trial.
- Insulin NPH + Human Soluble Insulin ± Metformin: Insulin NPH was administered subcutaneously in the thigh once daily at bedtime as basal insulin. Human Soluble insulin was injected in the abdominal area subcutaneously 30 minutes before each meal as bolus insulin. Metformin was given to subjects who were taking metformin before this trial.
Period: Overall Study
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Started | 29 | 29
Completed | 29 | 27
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] — Recorded at Visit 1 (screening visit), which was 1 week but no earlier than 2 weeks prior to randomisation.
  years | 57.6 (10.2) | 55.8 (9.8) | 56.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Recorded at Visit 1 (screening visit), which was 1 week but no earlier than 2 weeks prior to randomisation.
  Participants
    Female | 14 | 15 | 29
    Male | 15 | 14 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants] — Recorded at Visit 1 (screening visit), which was 1 week but no earlier than 2 weeks prior to randomisation.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 29 | 29 | 58
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] — Recorded at Visit 1 (screening visit), which was 1 week but no earlier than 2 weeks prior to randomisation.
  cm | 164.2 (8.5) | 164.2 (8.4) | 164.2 (8.4)
Weight [Mean (Standard Deviation); unit: kg] — Recorded at Visit 1 (screening visit), which was 1 week but no earlier than 2 weeks prior to randomisation.
  kg | 70.9 (13.1) | 66.5 (9.0) | 68.7 (11.4)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Recorded at Visit 1 (screening visit), which was 1 week but no earlier than 2 weeks prior to randomisation.
  kg/m^2 | 26.09 (3.13) | 24.63 (2.67) | 25.36 (2.98)
Pre-trial treatment of oral antidiabetic drug [Number; unit: participants]
  Acarbose | 9 | 10 | 19
  Gliclazide | 0 | 3 | 3
  Glimepiride | 2 | 4 | 6
  Metformin | 13 | 8 | 21
  Metformin hydrochloride | 2 | 3 | 5
  Repaglinide | 2 | 2 | 4
Pre-trial insulin treatment [Number; unit: participants]
  basal insulin (once daily) | 6 | 7 | 13
  premixed insulin (twice daily) | 23 | 22 | 45
Glycosylated haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] — Recorded at Visit 1 (screening visit), which was 1 week but no earlier than 2 weeks prior to randomisation.
  percentage of glycosylated haemoglobin | 8.76 (0.73) | 8.49 (0.76) | 8.62 (0.75)
Type 2 diabetes [Number; unit: participants] | 29 | 29 | 58
Duration of diagnosed diabetes [Mean (Standard Deviation); unit: years] | 10.23 (5.08) | 11.97 (7.14) | 11.10 (6.20)
Diabetes complications [Number; unit: participants]
  Diabetic complications | 13 | 15 | 28
  Diabetic retinopathy | 7 | 8 | 15
  Diabetic neuropathy | 10 | 11 | 21
  Diabetic Nephropathy | 4 | 3 | 7
  Macroangiopathy | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean 8-point Plasma Glucose (PG) After Two Weeks of Treatment
Description: Mean value of 8-point PG was the arithmetic mean of all 8 time-instant PG values of the 8-point PG profile.
Time Frame: Week 0, week 2
Population: Full analysis set using LOCF (Last Observation Carried Forward) included all randomised subject. The 2 subjects who withdrew after randomisation were excluded from the efficacy analyses.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Number analyzed (Participants) | 29 | 27
mmol/L | -2.84 (0.27) | -2.80 (0.28)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After Two Weeks of Treatment
Description: The FPG referred to pre-breakfast plasma glucose.
Time Frame: Week 0, week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Number analyzed (Participants) | 29 | 27
mmol/L | -2.22 (0.34) | -2.29 (0.35)

3. Secondary Outcome: Change From Baseline in Mean 2-hour Post Prandial Plasma Glucose (2hPPG) of 3 Meals After Two Weeks of Treatment
Description: The mean 2hPPG was derived from the 8-point PG profile as the mean value of the available 120 minutes after each meal.
Time Frame: Week 0, week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Number analyzed (Participants) | 29 | 27
mmol/L | -4.00 (0.39) | -3.47 (0.40)

4. Secondary Outcome: Change From Baseline in Mean Value of Pre-lunch, Pre-dinner and Bedtime PG After Two Weeks of Treatment
Description: The mean value of pre-lunch, pre-dinner and bedtime PG was derived from the 8-point PG profile measured before lunch, dinner and bedtime.
Time Frame: Week 0, week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Number analyzed (Participants) | 29 | 27
mmol/L | -2.47 (0.38) | -2.87 (0.38)

5. Secondary Outcome: Percentage of Subjects Achieving FPG < 6.0 mmol / L After Two Weeks of Treatment
Time Frame: Week 2
Population: Full analysis set using LOCF (Last Observation Carried Forward) included all randomised subject.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Number analyzed (Participants) | 29 | 29
percentage (%) of subjects | 48.3 | 48.3

6. Secondary Outcome: Percentage of Subjects Achieving Mean 2hPPG of 3 Meals < 8.0 mmol / L After Two Weeks of Treatment
Time Frame: Week 2
Population: Full analysis set using LOCF (Last Observation Carried Forward) included all randomised subject.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Number analyzed (Participants) | 29 | 29
percentage (%) of subjects | 41.4 | 34.5

7. Secondary Outcome: Percentage of Subjects Achieving Both FPG and 2hPPG Targets After Two Weeks of Treatment
Description: FPG target was < 6.0 mmol / L, 2hPPG target was < 8.0 mmol / L.
Time Frame: Week 2
Population: Full analysis set using LOCF (Last Observation Carried Forward) included all randomised subject.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Number analyzed (Participants) | 29 | 29
percentage (%) of subjects | 20.7 | 20.7

8. Secondary Outcome: Percentage of Subjects Achieving FPG Target Without Nocturnal Hypoglycaemia After Two Weeks of Treatment
Description: FPG target was < 6.0 mmol / L. Nocturnal hypoglycaemia was defined as a hypoglycaemic episode happened between 00:01 and 05:59 a.m. (both included).
Time Frame: Week 2
Population: Full analysis set using LOCF (Last Observation Carried Forward) included all randomised subject.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Number analyzed (Participants) | 29 | 29
percentage (%) of subjects | 41.4 | 34.5

9. Secondary Outcome: Change From Baseline in Fructosamine After Two Weeks of Treatment
Time Frame: Week 0, week 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Umol/L
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Number analyzed (Participants) | 29 | 27
Umol/L | -31.0 (5.37) | -23.7 (5.50)

10. Secondary Outcome: Incidence of Hypoglycaemic Episodes
Description: All events summarized were treatment emergent hypoglycaemic events. Hypoglycaemic episodes were summarized based on the ADA classification and also according to an additional definition.
  Severe hypoglycemia: ADA definition. Minor hypoglycaemic episode: an episode with symptoms with confirmation by plasma glucose (PG) < 3.1 mmol/l (56 mg/dl) and was handled by the subject himself/herself, or any asymptomatic PG value < 3.1 mmol/l (56 mg/dl).
  A hypoglycaemia episode was defined as nocturnal if the time of onset was between 00:01 and 05:59 a.m. (both included), otherwise it was diurnal.
Time Frame: Weeks 0-2
Population: Safety analysis set included all subjects receiving at least one dose of the trial products.
Measure: Number; unit: events
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Number analyzed (Participants) | 29 | 29
events
  All events | 22 | 54
  Severe | 0 | 0
  Nocturnal | 4 | 11
  Diurnal | 18 | 43
  Minor | 2 | 11

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timeframe of 2 weeks.
Description: Safety analysis set included all subjects receiving at least one dose of the trial products. All adverse events summarised were treatment emergent adverse events.
Arm/Group | Insulin Detemir + Insulin Aspart ± Metformin | Insulin NPH + Human Soluble Insulin ± Metformin
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 2/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir + Insulin Aspart ± Metformin (N=29) | Insulin NPH + Human Soluble Insulin ± Metformin (N=29)
upper restiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) — In the clinical trial report, the overall conclusion "No adverse event (AE) with incidence ≥ 5 % was reported in this trial" was based on treatment emergent AEs experienced by at least 5% of all subjects. The incidence in the total subjects was 3.4%.

LIMITATIONS AND CAVEATS:
The size of population analysed in study was smaller than that planned in the protocol. Therefore, the superiority of experimental products to comparator could not be concluded with sufficient statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones, for example, when the clinical trial report is available. At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.